CLINICAL TRIAL: NCT01961310
Title: Evaluation of the Intestinal Microbiota and Bacterial Translocation in Patients With Rheumatoid Arthritis
Acronym: MICROPOLY
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOIt/2012/JPL-01; 2014-A01753-44 (Other: ANSM)
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2020-07

CONDITIONS: Arthritis, Rheumatoid
Keywords: bacterial translocation; intestinal microbiota
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Bacterial Translocation; Occult Blood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RA patients: This group is composed of 25 patients with RA. The diagnosis of RA is based upon the American College of Rheumatology criteria.
  * Intervention: Plasma analysis for bacterial translocation
  * Intervention: Stool analysis
  Interventions: Biological: Plasma analysis for bacterial translocation; Biological: Stool analysis
- Healthy voluteers: This group is composed of 25 healthy volunteers.
  * Intervention: Plasma analysis for bacterial translocation
  * Intervention: Stool analysis
  Interventions: Biological: Plasma analysis for bacterial translocation; Biological: Stool analysis

INTERVENTIONS:
Biological: Plasma analysis for bacterial translocation — 1 ml of plasma will be obtained (blood sample). DNA will be extracted and amplified, and real-time quantitative PCR (polymerase chain reaction) performed.
Biological: Stool analysis — DNA from stool samples will be extracted, amplified, and used to identify the bacteria species present.

SUMMARY:
The main objective of this study is to compare the intestinal microbiota in newly diagnosed rheumatoid arthritis (RA) with that from individuals without RA.

The first analysis will compare the proportion of filamentous bacteria in the intestinal microbiota between the two groups.

DETAILED DESCRIPTION:
The secondary objectives of this study are :

* A. To compare between the two groups :
* a. The proportion of Proteus mirabilis in the intestinal microbiota;
* b . The proportion of species producing peptidyl arginine deaminase (PAD ) in the intestinal microbiota;
* c . The number of species found in the intestinal microbiota.
* B. To evaluate bacterial translocation (from the digestive tract) in newly diagnosed RA patients with and healthy volunteers without RA. (Bacterial translocation is a phenomenon in which live bacteria or a part of bacteria (e.g. LPS teichoïc acid) cross the intestinal barrier and reach the bloodstream.).
* C. To describe the ecology of the intestinal microbiota of newly diagnosed RA patients (characterization of species found according to their respiratory metabolism, according to their bacteriological characteristics, and according to whether or not the species are found significantly more frequently in patients with RA than in individuals without RA).

ELIGIBILITY:
Inclusion Criteria for RA patients:

* The patient was correctly informed
* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* No antibiotic treatments within the 30 days preceding inclusion
* Absence of digestive pathology
* RA diagnosis made within the past 12 months

Exclusion Criteria for RA patients:

* The patient has participated in another study within the past 3 months
* The patient is under judicial protection, or any kind of guardianship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient has taken antibiotics in the 30 days preceding inclusion
* RA was diagnosed more than 12 months ago
* Digestive pathology

Inclusion Criteria for healthy volunteers (HV):

* The HV was correctly informed
* The HV must have given his/her informed and signed consent
* The HV must be insured or beneficiary of a health insurance plan
* Absence of digestive pathology
* No antibiotic treatments within the 30 days preceding inclusion
* Does not have RA

Exclusion Criteria for HVs:

* The HV has participated in another study within the past 3 months
* The HV is under judicial protection, or any kind of guardianship
* The HV refuses to sign the consent
* It is impossible to correctly inform the HV
* The HV is pregnant, parturient, or breastfeeding
* The HV has taken antibiotics in the 30 days preceding inclusion
* Digestive pathology
* Joint pathology of any kind (including inflammatory pathologies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 50 adult subjects will be included: 25 with newly diagnosed RA (<12 months) based on the American College of Rheumatology criteria, and 25 healthy volunteers without RA.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
The proportion of filamentous bacteria in the intestinal microbiota | Baseline (day 0)

SECONDARY OUTCOMES:
The proportion of Proteus mirabilis in the intestinal microbiota | baseline (Day 0)
The proportion of species producing peptidyl arginine desaminase (PAD) in the intestinal microbiota | baseline (Day 0)
The number of species found in the intestinal microbiota | baseline (Day 0)
Presence/absence of bacterial translocation | baseline (Day 0)
Description of the ecology of intestinal microbiota | baseline (Day 0)
  Diversity indices according to species and/or functional groups. The general goal is to provide a description of the functional differences between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Dunyach-Rempy, PharmD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes; Jean Philippe Lavigne, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - CHRU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - Unité U1047 "Bacterial virulence and infectious diseases", UFR de Médecine, Nîmes

REFERENCES:
- [Result] Dunyach-Remy C, Pouget C, Pers YM, Gaujoux-Viala C, Demattei C, Salipante F, Grenga L, Armengaud J, Lavigne JP, Jorgensen C. Participation of gut microbiota and bacterial translocation in chronic systemic inflammation in recently diagnosed rheumatoid arthritis patients. Curr Res Microb Sci. 2025 Feb 24;8:100366. doi: 10.1016/j.crmicr.2025.100366. eCollection 2025. PMID 40123592